CLINICAL TRIAL: NCT02359695
Title: Low-dose Growth Hormone Supplementation Increases Clinical Pregnancy Rate in Poor Responders Undergoing in Vitro Fertilisation.
Brief Title: Low-dose GH Supplementation Increases Clinical Pregnancy Rate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centro de Infertilidad y Reproducción Humana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIRH-BROHC-2013; 2013-003123-11 (EudraCT Number)
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Infertility
Keywords: Poor ovarian response; IVF; Growth hormone
MeSH Terms: conditions — Infertility | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GH cycle (Experimental): Subsequent IVF cycle, supplemented with a low dose of growth hormone.
  Interventions: Drug: Growth Hormone

INTERVENTIONS:
Drug: Growth Hormone — A dose of 0.5 IU of growth hormone will be administered daily from the first day of the agonist until the day of hCG administration
  Other Names: Somatotropin

SUMMARY:
The objective of this study is to assess whether a low dose of GH supplementation (0.5 IU/day) increases clinical pregnancy rates in women with a history of POR who failed to become pregnant in two previous IVF cycles.

DETAILED DESCRIPTION:
The investigators aim to study the impact of a low-dose growth hormone (GH) supplementation in pregnancy rates in poor responders in a prospective, self-controlled study of 64 poor responders to previous IVF cycles who failed to achieve pregnancy and were supplemented with low-doses of GH in a subsequent cycle using the same gonadotropin dose and protocol. Our primary endpoint was the clinical pregnancy rate (CPR), considering secondary endpoints the number of retrieved oocytes, embryos, embryo quality and the proportion of cycles with embryo transfer.

Controlled ovarian hyperstimulation will be performed using a GnRH agonist long protocol from day 21-23 of the menstrual cycle at a dose of 1 mg/ day, using the same schedule and dose as in the previous cycle, so that the only difference between them is the GH supplementation.

After confirming pituitary inhibition, the dose of GnRH agonist will be decreased to 0.5 mg/day, and COH will begin with gonadotropins at a dose of 300 UI, subsequently adjusting according to clinical response. Human chorionic gonadotropin (hCG) will be administered when follicles reached > 17 mm in diameter. A dose of 0.5 IU of GH will be administered daily from the first day of the agonist until the day of hCG administration. Oocyte retrieval will be performed 36 hours after hCG administration by ultrasound-guided follicle aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of POR, defined according to the Bologna criteria
* Absence of pregnancy in at least two previous IVF cycles

Exclusion Criteria:

* Body mass index ≥ 30 kg/m2
* Presence of endocrinopathies
* Altered karyotype in one or both partners
* History of invasive ovarian surgery
* History of chronic, autoimmune or metabolic diseases
* Altered meiosis in testicular biopsy or altered sperm-FISH
* Drug therapy in the male partner
* Participation, within the previous 6 months, in another clinical trial with medication

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 7 weeks of gestation
  Presence of an intrauterine gestational sac with embryonic cardiac activity display, evaluated by ultrasound

SECONDARY OUTCOMES:
Retrieved oocytes | On egg retrieval day
  Total number of retrieved oocytes
Number of obtained embryos | 3 days after egg retrieval
  Total number of obtained embryos
Embryo quality | 3 days after embryo transfer
  Total number of top quality embryos per cycle
Proportion of cycles with embryo transfer | 3 days after egg retrieval
  Proportion of cycles reaching embryo transfer per initiated cycle

CONTACTS AND LOCATIONS:
Overall Officials: Mario Brassesco, MD, Study Director — Centro de Infertilidad y Reproducción Humana
Locations (1):
- Centro de Infertilidad y Reproducción Humana (CIRH), Barcelona, Spain